## APPROVED BY THE YALE UNIVERSITY IRB 10/23/2019 NCT03089983

## MEDICAL ETHICS COMMITTEE UNIVERSITY MALAYA MEDICAL CENTRE

## CONSENT BY PATIENT FOR CLINICAL RESEARCH

**Version No.:** 4

Version Date: April 18, 2018

| I, | | (Name of Patient) |
|---|---|---|
| Identity Card No | in | (Address) |
| hereby agree to take part in the clinical research (clinical study/questionnaire study/drug trial) specified | | |
| below: | | |
| Title of Study: Addiction, HIV and Tuber | rculosis in Malaysian Criminal Justi | ce Settings |
| Aim 1b: A Randomized Control Trial to Compare Completion Rates and Tolerability of Standard vs<br>Short-course Latent Tuberculosis Infection Treatment among Prisoners in Malaysia | | |
| The nature and purpose of which has been explained to me by | | |
| | (. | Name of Research staff) |
| and interpreted by | (Name & Desig | gnation of Interpreter) |
| to the best of his/her ability in | language/dialect. | |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. | | |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. | | |
| Date: | Signature(Subject patie | |

## APPROVED BY THE YALE UNIVERSITY IRB 10/23/2019

| IN THE PRESENCE OF |
|---|
| Name |
| Identity Card No. |
| Signature(Witness for Signature of Patient) |
| Designation |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. |
| Signature Date |

| CONSENT BY PATIENT FOR CLINICAL RESEARCH |
|------------------------------------------|
| IC NO. |
| SUBJECT ID. |
| NAME |
| SEX |
| AGE |

BK-MIS-1117-E02